CLINICAL TRIAL: NCT04992481
Title: Influence of Fluoride Varnish, Ozone and Octenidin on the Incidence of White Spot Lesions and Caries During Orthodontic Treatment - a Randomized Clinical Trial
Brief Title: Fluoride Varnish, Ozone, Octenidin and WSLs in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Katarzyna Grocholewicz, Professor, Pomeranian Medical University Szczecin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KB-0012/124/12
Record Dates: First submitted 2021-07-19; First posted 2021-08-05 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: White Spot Lesion of Tooth
Keywords: white spot; orthodontic treatment; caries prophylaxis

STUDY DESIGN:
Intervention Model Description: To participate in the study 167 healthy adults (16-50 years) who began orthodontic treatment with fixed appliances bonded to both dental arches were eligible and consecutively invited. Informed consent was obtained from 150 patients (111 women and 39 men). The patients have been randomly divided (using number random generator) into five groups (n=30), including four study groups (I, II, III, IV) and one control group (K).
Who Masked: Investigator
Masking Description: The patients have been randomly divided (using number random generator) into five groups (n=30), including four study groups (I, II, III, IV) and one control group (K).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1. professional mechanical tooth cleaning (PMTC)+fluoride varnish (Experimental): This arm constituted of randomly selected 30 participants. In this group professional mechanical tooth cleaning (PMTC)+fluoride varnish were performed.
  Interventions: Procedure: PMTC; Procedure: fluoride varnish
- 2. PMTC+fluoride varnish+gaseous ozone therapy (Experimental): This arm constituted of randomly selected 30 participants. In this group PMTC+fluoride varnish+gaseous ozone therapy were performed.
  Interventions: Procedure: PMTC; Procedure: fluoride varnish; Procedure: gaseous ozone therapy
- 3. PMTC+fluoride varnish+domestic octenidin mouth rinse (Experimental): This arm contituted of randomly selected 30 participants. In this group PMTC+fluoride varnish+domestic octenidin mouth rinse were applied.
  Interventions: Procedure: PMTC; Procedure: fluoride varnish; Procedure: domestic octenidin mouth rinse
- 4. PMTC+fluoride varnish+domestic octenidin mouth rinse+ gaseous ozone therapy (Experimental): This arm constituted of randomly selected 30 participants. In this group PMTC+fluoride varnish+domestic octenidin mouth rinse+ gaseous ozone therapy were performed.
  Interventions: Procedure: PMTC; Procedure: fluoride varnish; Procedure: gaseous ozone therapy; Procedure: domestic octenidin mouth rinse
- Control group (No Intervention): Control group not subjected to any prophylactic program constituted of randomly selected 30 participants.

INTERVENTIONS:
Procedure: PMTC — In patients from the study groups I, II, III, IV a professional mechanical tooth cleaning (PMTC) including air-polishing was proceeded on every visit using a glycine-based prophylaxis powder (Air-Flow Soft, EMS, Switzerland).
  Arms: 1. professional mechanical tooth cleaning (PMTC)+fluoride varnish; 2. PMTC+fluoride varnish+gaseous ozone therapy; 3. PMTC+fluoride varnish+domestic octenidin mouth rinse; 4. PMTC+fluoride varnish+domestic octenidin mouth rinse+ gaseous ozone therapy
Procedure: fluoride varnish — In patients from groups I, II, III, IV a fluoride varnish of 5% NaF (Profluorid Varnish, Voco, Germany) was applied with a microbrush. Every patient was instructed to stop from drinking and eating for the next two hours (as recommended by the manufacturer).
  Arms: 1. professional mechanical tooth cleaning (PMTC)+fluoride varnish; 2. PMTC+fluoride varnish+gaseous ozone therapy; 3. PMTC+fluoride varnish+domestic octenidin mouth rinse; 4. PMTC+fluoride varnish+domestic octenidin mouth rinse+ gaseous ozone therapy
Procedure: gaseous ozone therapy — Patients from groups II and IV were additionally subjected to in-office ozone therapy using OzonyTron-OZ (Mymed, Germany). Ozone was applied on a silicone double-jaw tray of a proper size (allowing even ozone distribution in the oral cavity) following professional mechanical tooth cleaning. A Full Mouth Desinfection program lasting 5 minutes was used.
  Arms: 2. PMTC+fluoride varnish+gaseous ozone therapy; 4. PMTC+fluoride varnish+domestic octenidin mouth rinse+ gaseous ozone therapy
Procedure: domestic octenidin mouth rinse — Patients from groups III and IV received a domestic mouthrinse (Octenidol MD, Schülke, Germany) and were recommended to use 15 ml of the liquid for 30 seconds after evening toothbrushing.
  Arms: 3. PMTC+fluoride varnish+domestic octenidin mouth rinse; 4. PMTC+fluoride varnish+domestic octenidin mouth rinse+ gaseous ozone therapy

SUMMARY:
Objectives: to assess the efficiency of four prophylactic protocols on white spot lesions during orthodontic treatment: 1. professional mechanical tooth cleaning (PMTC)+fluoride varnish, 2. PMTC+fluoride varnish+gaseous ozone therapy 3. PMTC+fluoride varnish+domestic octenidin mouth rinse, 4. PMTC+fluoride varnish+domestic octenidin mouth rinse+ gaseous ozone therapy versus a control group not subjected to any prophylactic program.

Materials and Methods: Patients (n=150, 111 women and 39 men, age 16-50y,) who began orthodontic treatment with fixed appliances bonded to both dental arches have been provided with detailed initial oral hygiene instruction recommendations. The hygienic recommendations comprised: toothbrushing every surface after every meal (4 minutes) with a fluoridated toothpaste (1450 ppm) using the roll and Bass methods with a soft toothbrush recommended for fixed appliance, interdental toothbrushes, single-tufted brushes and dental floss recommended for fixed appliance. An instruction leaflet has been delivered to every subject, as well. A reinstruction was made during every control visit referring to the results of the oral hygiene assessment.

Subsequently, the patients were randomly allocated (using number random generator) into five groups (n=30), including four study groups (I, II, III, IV) and one control group (K). Group I: professional mechanical tooth cleaning (PMTC)+fluoride varnish, group II: PMTC+fluoride varnish+gaseous ozone therapy, group III: PMTC+fluoride varnish+domestic octenidin mouth rinse, group IV: PMTC+fluoride varnish+domestic octenidin mouth rinse+ gaseous ozone therapy, control group (K) not subjected to any prophylactic program.

The period of observation was 12 months, with prophylactic visits every four weeks and examinations every 12 weeks. The assessment of white spot lesions was proceeded on the labial surfaces of upper and lower teeth, with patient on the dental chair in proper dental lighting, after cleaning and drying the assessed surfaces.

DETAILED DESCRIPTION:
In the recent years orthodontic treatment has become very popular. Patients seek orthodontic treatment, mainly to improve the esthetics of their smiles, since appearance has become extremely important in the modern society. Another reason to have orthodontic treatment is striving for a better, more comfortable occlusion. However, complications of orthodontic therapy may occur.

Bonding an orthodontic appliance creates environment for bacterial adhesion, with reduced salivary flow. The most retentive sites are: area between the bracket upper surface and gingival margin as well as proximal surfaces. The resulting pH reduction in this area promotes the demineralization process. Enamel demineralization, being an initial stage of caries as well as gingival inflammation belong to the most prevalent detrimental effects resulting from increased accumulation of the biofilm and difficulty to clean these surfaces.

With treatment initiation the microbial environment of the oral cavity changes - increases the number of Lactobacillus and Streptococcus mutans in biofilm.

White spot lesions (WSLs) are the first sings of carious lesions on enamel that can be detected with the naked eye and result from demineralization. WSLs may arise as early as four or even two weeks following bonding fixed appliance creating a need for a clinical intervention.

The most often affected teeth are lateral incisors, followed by canines, premolars and central incisors. There is no side predilection, or difference for upper and lower dental arches. At least one new initial carious lesion is found in 72,9% patients, whereas in 61% cavities develop during the first twelve months of orthodontic treatment. A fast increase of the incidence of WSLs is observed during the first six months of treatment - initial caries is found in 38% patients, after 12 months WSLs are found in 46% patients.

Caries prevention in patients under orthodontic treatment is based on hygienic regimen, in order to prevent biofilm accumulation by proper brushing technique, use of fluoride, as well as bactericidal chemicals, including chlorhexidine, octenidin, ozone, casein phosphopeptides-amorphous calcium phosphate (CPP-ACP).

The alterations of enamel structure within WSLs are only partially reversible. The number of WSLs does not return to that from before orthodontic treatment even 12 years after debonding. The treatment methods comprise: remineralization (with fluoride or hydroxyapatite), resin infiltration, microabrasion, restorative treatment or veneers, depending on the severity of the destruction .

WSLs constitute a health and an esthetic problem thus introducing preventive measures and early detection of WSLs is essential. A patient prepared for orthodontic treatment should be aware of the need for a high hygienic regimen.

In patients with increased caries risk professional fluoride prophylaxis, using a varnish or gel should be considered. In-office application of fluoride varnish allows for better control of application and is independent from patient's domestic cooperation. A meta-analysis research based on 36 RCTs showed that NaF varnish is the most effective agent in the prevention of orthodontically induced WSLs. Application of fluoride varnish on every orthodontic appointment reduces enamel demineralization by 44% comparing to placebo.

Ozone is a strong oxidant, destructing to pathogens; exerts bactericidal, antiviral and fungicidal activity as well as stimulates tissue metabolism by increasing oxidation. It reduces inflammation, by stimulating interleukin and interferon production, enables remineralization, breaking protein chains and oxidating aminoacids.

Octenidin dihydrochloride exerts antimicrobial action on: S. mutans, Str. sanguis, A. viscosus, A. naeslundii, influencing the biofilm.

Study goals and objectives The aim of the present study was to assess the efficiency of four prophylactic protocols on white spot lesions during orthodontic treatment: 1. professional mechanical tooth cleaning (PMTC)+fluoride varnish, 2. PMTC+fluoride varnish+gaseous ozone therapy 3. PMTC+fluoride varnish+domestic octenidin mouth rinse, 4. PMTC+fluoride varnish+domestic octenidin mouth rinse+ gaseous ozone therapy versus a control group not subjected to any prophylactic program.

Study Design The study was conducted in years 2013-2016 in 150 participants (111 females and 39 males) aged from 16 to 50 years, who were recruited from a pool of patients attending Department of Interdisciplinary Dentistry at Pomeranian Medical University in Szczecin, Poland. The study protocol was approved by the Ethics Committee of the Pomeranian Medical University in Szczecin (KB-0012/124/12) and conducted in accordance with accepted ethical standards for research practice. A written informed consent was obtained from all participants enrolled. The study protocol has been registered in clinicaltrials.gov (reference number NCT04147091).

Methodology Sample size calculation for repeated-measures ANOVA was performed by using the R function wp.rmanova, WebPower package. The power of correlation was established at the level of 0,75.

To participate in the study 167 healthy adults (16-50 years) who began orthodontic treatment with fixed appliances bonded to both dental arches were eligible and consecutively invited. Informed consent was obtained from 150 patients (111 women and 39 men). The patients have been randomly divided (using number random generator) into five groups (n=30), including four study groups (I, II, III, IV) and one control group (K).

Detailed initial oral hygiene instruction recommendations have been provided to every patient. The hygienic recommendations comprised: toothbrushing every surface after every meal (4 minutes) with a fluoridated toothpaste (1450 ppm) using the roll and Bass methods with a soft toothbrush recommended for fixed appliance, interdental toothbrushes, single-tufted brushes and dental floss recommended for fixed appliance. An instruction leaflet has been delivered to every subject, as well. A reinstruction was made during every control visit referring to the results of the oral hygiene assessment.

The distribution of prophylaxis procedures (performed every four weeks) in the study and control groups has been presented in Consort flow diagram. In patients from the study groups I, II, III, IV a professional mechanical tooth cleaning (PMTC) including air-polishing was proceeded on every visit using a glycine-based prophylaxis powder (Air-Flow Soft, EMS, Switzerland).

In patients from groups I, II, III, IV a fluoride varnish of 5% NaF (Profluorid Varnish, Voco, Germany) was applied with a microbrush. Every patient was instructed to stop from drinking and eating for the next two hours (as recommended by the manufacturer).

Patients from groups II and IV were additionally subjected to in-office ozone therapy using OzonyTron-OZ (Mymed, Germany). Ozone was applied on a silicone double-jaw tray of a proper size (allowing even ozone distribution in the oral cavity) following professional mechanical tooth cleaning. A Full Mouth Desinfection program lasting 5 minutes was used.

Patients from groups III and IV received a domestic mouthrinse (Octenidol MD, Schülke, Germany) and were recommended to use 15 ml of the liquid for 30 seconds after evening toothbrushing.

Patients assigned to control group had no professional hygienic or prophylactic procedures performed, despite for initial oral hygiene instruction and written dietetic recommendations.

The period of observation was 12 months, with prophylactic visits every four weeks and examinations every 12 weeks. The assessment of white spot lesions was proceeded on the labial surfaces of upper and lower teeth, with patient on the dental chair in proper dental lighting, after cleaning and drying the assessed surfaces. WSL index according to Gorelick et al. was used as follows:

0 - no visible WSL or surface disruption (no demineralization)

1. - visible WSL, covering less than 1/3 of surface, without surface disruption (mild demineralization)
2. - visible WSL, covering more than 1/3 of the surface, with a roughened surface, but not requiring restoration (moderate demineralization)
3. - visible cavitation, requiring restoration (severe demineralization) Every dental surface was subjected to visual-tactile examination performed on a dental chair with proper dental lighting, using dental probe and a mirror. Caries was diagnosed on the level of cavitation, the presence of fillings has been noted as well.

Follow-Up This study has a 1-year follow-up.

Data Management and Statistical Analysis All continuous variables were verified for distribution normality using Kołmogorov-Smirnov test, ShapiroWilk test, also by qqplots. Statistical significance of differences between two groups were analyzed using Student t-test and Mann-Whitney test and between multiple groups - analysis of variance (ANOVA), Tukey HSD test or Kruskal-Wallis test.

Discontinuous variables were described by their number and frequency of occurrence. Statistical correlations between discontinuous variables were analyzed using χ2 Pearson's test or exact Fisher's test.

For the study of correlations between discontinuous variables: ordinal and nominal (coded variables: 0/1) and continuous variables rank Spearman correlation coefficient was used. The results have been described using the correlation coefficient r and the level of significance p.

All statistical analyzes with data visualization have been programmed in the interpreted programming language "R" with open-source software for data science, scientific research, and technical communication "R studio" version 1.4.1106. The level p=0,051-0,099 has been set as a borderline trend of statistical significance. Computer software STATA 11 (2009) of license No 30110532736 has been used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

* permanent dentition
* fixed appliances bonded to both dental arches (no more than 4 weeks prior to the study)

Exclusion Criteria:

* inborn tooth anormalities
* prosthetics restorations

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
WSLs presence on teeth | 12 months
  The assessment of white spot lesions was proceeded on the labial surfaces of upper and lower teeth, with patient on the dental chair in proper dental lighting, after cleaning and drying the assessed surfaces. WSL index according to Gorelick et al. [28] was used as follows:
  0 - no visible WSL or surface disruption (no demineralization)
  * visible WSL, covering less than 1/3 of surface, without surface disruption (mild demineralization)
  * visible WSL, covering more than 1/3 of the surface, with a roughened surface, but not requiring restoration (moderate demineralization)
  * visible cavitation, requiring restoration (severe demineralization) Every dental surface was subjected to visual-tactile examination performed on a dental chair with proper dental lighting, using dental probe and a mirror. Caries was diagnosed on the level of cavitation, the presence of fillings has been noted as well.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Grocholewicz, DDS, PhD, Study Chair — Pomeranian Medical University, Szczecin, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Øgaard B: White spot lesions during orthodontic treatment: mechanisms and fluoride preventive aspects. Semin Orthod. 2008;14:183-193
- [Result] Scheie AA, Arneberg P, Krogstad O. Effect of orthodontic treatment on prevalence of Streptococcus mutans in plaque and saliva. Scand J Dent Res. 1984 Jun;92(3):211-7. doi: 10.1111/j.1600-0722.1984.tb00881.x. PMID 6589736
- [Result] Fejerskov O, Nyvad B, Kidd E: Clinical and histological manifestations of dental caries. In: Fejerskov O, Kidd E, editors. Dental caries: the disease and its clinical management. Copenhagen, Denmark: Blackwell Munksgaard; 2003, p. 71-99.
- [Result] Ogaard B, Rolla G, Arends J. Orthodontic appliances and enamel demineralization. Part 1. Lesion development. Am J Orthod Dentofacial Orthop. 1988 Jul;94(1):68-73. doi: 10.1016/0889-5406(88)90453-2. PMID 3164585
- [Result] Tufekci E, Dixon JS, Gunsolley JC, Lindauer SJ. Prevalence of white spot lesions during orthodontic treatment with fixed appliances. Angle Orthod. 2011 Mar;81(2):206-10. doi: 10.2319/051710-262.1. PMID 21208070
- [Result] Shungin D, Olsson AI, Persson M. Orthodontic treatment-related white spot lesions: a 14-year prospective quantitative follow-up, including bonding material assessment. Am J Orthod Dentofacial Orthop. 2010 Aug;138(2):136.e1-8; discussion 136-7. doi: 10.1016/j.ajodo.2009.05.020. PMID 20691346
- [Result] Kozak U, Sekowska A, Chalas R. The Effect of Regime Oral-Hygiene Intervention on the Incidence of New White Spot Lesions in Teenagers Treated with Fixed Orthodontic Appliances. Int J Environ Res Public Health. 2020 Dec 17;17(24):9460. doi: 10.3390/ijerph17249460. PMID 33348756
- [Result] Chapman JA, Roberts WE, Eckert GJ, Kula KS, Gonzalez-Cabezas C. Risk factors for incidence and severity of white spot lesions during treatment with fixed orthodontic appliances. Am J Orthod Dentofacial Orthop. 2010 Aug;138(2):188-94. doi: 10.1016/j.ajodo.2008.10.019. PMID 20691360
- [Result] Maxfield BJ, Hamdan AM, Tufekci E, Shroff B, Best AM, Lindauer SJ. Development of white spot lesions during orthodontic treatment: perceptions of patients, parents, orthodontists, and general dentists. Am J Orthod Dentofacial Orthop. 2012 Mar;141(3):337-344. doi: 10.1016/j.ajodo.2011.08.024. PMID 22381494
- [Result] Derks A, Kuijpers-Jagtman AM, Frencken JE, Van't Hof MA, Katsaros C. Caries preventive measures used in orthodontic practices: an evidence-based decision? Am J Orthod Dentofacial Orthop. 2007 Aug;132(2):165-70. doi: 10.1016/j.ajodo.2005.10.028. PMID 17693365
- [Result] Stecksen-Blicks C, Renfors G, Oscarson ND, Bergstrand F, Twetman S. Caries-preventive effectiveness of a fluoride varnish: a randomized controlled trial in adolescents with fixed orthodontic appliances. Caries Res. 2007;41(6):455-9. doi: 10.1159/000107932. Epub 2007 Sep 7. PMID 17827963
- [Result] Ogaard B, Larsson E, Henriksson T, Birkhed D, Bishara SE. Effects of combined application of antimicrobial and fluoride varnishes in orthodontic patients. Am J Orthod Dentofacial Orthop. 2001 Jul;120(1):28-35. doi: 10.1067/mod.2001.114644. PMID 11455374
- [Result] Geiger AM, Gorelick L, Gwinnett AJ, Benson BJ. Reducing white spot lesions in orthodontic populations with fluoride rinsing. Am J Orthod Dentofacial Orthop. 1992 May;101(5):403-7. doi: 10.1016/0889-5406(92)70112-N. PMID 1590288
- [Result] Demito CF, Vivaldi-Rodrigues G, Ramos AL, Bowman SJ. The efficacy of a fluoride varnish in reducing enamel demineralization adjacent to orthodontic brackets: an in vitro study. Orthod Craniofac Res. 2004 Nov;7(4):205-10. doi: 10.1111/j.1601-6343.2004.00305.x. PMID 15562583
- [Result] Msallam FA, Grawish ME, Hafez AM, Abdelnaby YL. Decalcification prevention around orthodontic brackets bonded to bleached enamel using different topical agents. Prog Orthod. 2017 Dec;18(1):15. doi: 10.1186/s40510-017-0170-4. Epub 2017 Jun 12. PMID 28580541
- [Result] Sharda S, Gupta A, Goyal A, Gauba K. Remineralization potential and caries preventive efficacy of CPP-ACP/Xylitol/Ozone/Bioactive glass and topical fluoride combined therapy versus fluoride mono-therapy - a systematic review and meta-analysis. Acta Odontol Scand. 2021 Aug;79(6):402-417. doi: 10.1080/00016357.2020.1869827. Epub 2021 Jan 16. PMID 33459095
- [Result] Hochli D, Hersberger-Zurfluh M, Papageorgiou SN, Eliades T. Interventions for orthodontically induced white spot lesions: a systematic review and meta-analysis. Eur J Orthod. 2017 Apr 1;39(2):122-133. doi: 10.1093/ejo/cjw065. PMID 27907894
- [Result] Tahmasbi S, Mousavi S, Behroozibakhsh M, Badiee M. Prevention of white spot lesions using three remineralizing agents: An in vitro comparative study. J Dent Res Dent Clin Dent Prospects. 2019 Winter;13(1):36-42. doi: 10.15171/joddd.2019.006. Epub 2019 Apr 24. PMID 31217917
- [Result] Lale S, Solak H, Hincal E, Vahdettin L. In Vitro Comparison of Fluoride, Magnesium, and Calcium Phosphate Materials on Prevention of White Spot Lesions around Orthodontic Brackets. Biomed Res Int. 2020 Mar 30;2020:1989817. doi: 10.1155/2020/1989817. eCollection 2020. PMID 32337230
- [Result] Hu H, Feng C, Jiang Z, Wang L, Shrestha S, Yan J, Shu Y, Ge L, Lai W, Hua F, Long H. Effectiveness of remineralizing agents in the prevention and reversal of orthodontically induced white spot lesions: a systematic review and network meta-analysis. Clin Oral Investig. 2020 Dec;24(12):4153-4167. doi: 10.1007/s00784-020-03610-z. Epub 2020 Oct 15. PMID 33057826
- [Result] Gorelick L, Geiger AM, Gwinnett AJ. Incidence of white spot formation after bonding and banding. Am J Orthod. 1982 Feb;81(2):93-8. doi: 10.1016/0002-9416(82)90032-x. PMID 6758594
- [Derived] Grocholewicz K, Miklasz P, Zawislak A, Sobolewska E, Janiszewska-Olszowska J. Fluoride varnish, ozone and octenidine reduce the incidence of white spot lesions and caries during orthodontic treatment: randomized controlled trial. Sci Rep. 2022 Aug 17;12(1):13985. doi: 10.1038/s41598-022-18107-w. PMID 35978074